CLINICAL TRIAL: NCT02800577
Title: An Exploratory Investigation in Depressed Patients Initiating Treatment With Citalopram, to Determine the Sensitivity and Specificity of the P1vital® Oxford GP-Emotional Test Battery in Predicting Drug Response and Non-response
Brief Title: Using Computer Tasks to Predict Response to Antidepressants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: P1vital Products Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1V-DEP-MD01
Record Dates: First submitted 2016-03-16; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All participants (Other): Study has a single, non-interventional arm where the General Practitioner Emotional Test Battery (GP-ETB) will be administered.
  Interventions: Device: General Practitioner Emotional Test Battery (GP-ETB)

INTERVENTIONS:
Device: General Practitioner Emotional Test Battery (GP-ETB) — The GP-ETB (Class I Medical Device) comprises three computer tasks. In the first task, the 'Emotional Categorisation Task' patients are given forty words that might be used to describe them and indicate whether they would 'like' or 'dislike' to be described by a particular word. In the 'Facial Expression Recognition Task' patients are asked to judge whether a briefly displayed face is expressing one of six emotions. In the final task, the 'Emotional Recall Task', the patient should recall as many words as they can from the series of words that were presented in the first task. The patients perform these tasks once before antidepressant treatment and again seven days after treatment begins.

SUMMARY:
In England over 800,000 patients each year are either newly diagnosed with depression or present with a new episode of depression in primary care. The majority of patients do not respond to the first drug prescribed and have to try several different antidepressants before an effective treatment is found. Antidepressants have a slow clinical onset of action, taking 4 to 6 weeks before changes in mood become apparent. No test exists to guide General Practitioners (GPs) as to whether their patient is responding to the prescribed successive treatments. This often results in delays of many months before patients return to good mental health. The GP-ETB is a set of computer-based emotional processing tasks. It was developed and optimised to be sensitive to early changes in emotional bias that are indicative of successful antidepressant treatment. The current investigation is an exploratory study using the GP-ETB.

It will test the predictive ability of the GP-ETB with regard to later subjective drug response and nonresponse. The study will recruit depressed patients from primary care settings. There are no study drugs prescribed as part of this clinical investigation. Eligible patients will have been prescribed citalopram by their GP prior to study entry. The decision to initiate treatment with citalopram will be independent of study participation. The duration of the study is 5 months. Each patient will be required to attend 3 visits and total duration of the study for the patient will be 46 weeks. During the visits patients will be asked to complete a variety of questionnaires and GP-ETB tasks on the computer. Sensitivity and specificity data collected during this study will be used to develop a computer algorithm intended to predict response at 46 weeks, based on GP-ETB data collected 1 week after initiation of antidepressant treatment.

DETAILED DESCRIPTION:
The study is an exploratory, single arm, multi-centre, clinical investigation of a medical device. The study consists of a recruitment period followed within 3 days by the first study visit. After a GP has decided to prescribe citalopram for depression, GP assesses patient for suitability for study and provides a brief explanation of study to potentially suitable patient. Patient signs pre-study consent form agreeing to being contacted by researcher from the same or another GP surgery and agreeing not to take their first dose of citalopram until after their first study visit.

Recruitment and pre-screening Main study Patient Information Sheet/Informed Consent Form (PIS/ICF) will be provided. Researcher will contact patient and book the Visit 1 within 3 days from GP visit.

At Visit 1, patients will be screened and eligible patients will be enrolled in the study. Visit 1 procedures include:

* Informed Consent
* Demographics
* Review of other medication
* Brief medical history including depression history (if applicable)
* Entry criteria check and enrolment into study
* Quick Inventory of Depressive Symptomatology Self Report (QIDS-SR)
* Montgomery-Åsberg Depression Rating Scale (MADRS)
* Beck Depression Inventory®II (BDI-II)
* GP-ETB (set of computer tasks)
* Review of Adverse Events (AEs) and Adverse Device Effects (ADEs) and device deficiencies Patients will return approximately 1 week later for Visit 2 and will complete a variety of questionnaires and assessments:
* QIDS-SR
* BDI-II
* GP-ETB
* Assessment of compliance with study prohibitions and restrictions
* Changes to antidepressant medication since last visit (e.g. increased dose, change of drug)
* Concordance with prescribed antidepressant medication, as determined through interview with patient
* Review of other medication
* Review of AEs, ADEs and device deficiencies Visit 3 will be scheduled to take place 46 weeks after the first dose of citalopram. The following questionnaires and assessments will be completed:
* QIDS-SR
* MADRS
* BDI-II
* Acceptability questionnaire(s) relating to use of GP-ETB (patient and researcher)
* Assessment of compliance with study prohibitions and restrictions
* Changes to antidepressant medication since last visit (e.g. increased dose, change of drug)
* Concordance with prescribed antidepressant medication, as determined through interview with patient
* Review of other medication
* Review of AEs, ADEs and device deficiencies At the end of the visit, patients will be considered to have completed the study.

Emotional Test Battery (GP-ETB) tasks: The GP-ETB is a series of computerised tasks during which participants must respond by button press to pictures (e.g. pictures of faces) or words presented on the screen. Some of the pictures are mildly emotional (e.g. a fearful face). Response bias for each Participant choice and reaction times are measured during the following tasks: Emotional Categorisation Task (ECAT) Number of words categorised as liked and disliked

% accuracy for each condition, Reaction time for each condition Emotional Recall Task (EREC) Total number of words recalled for each valence (positive, negative) Number of commission errors

Facial Expression Recognition Task (FERT):

* accuracy of recognition of each emotion (happiness, fear, anger, disgust, surprise, sadness, neutral)
* mis-classifications for each emotion Individual average reaction time for correct answers in each emotion Reaction time for all emotions Target sensitivity for each emotion Response bias for each emotion Questionnaires and rating scales: The questionnaires and rating scales used in the current study, except the acceptability questionnaires relating to use of GP-ETB (patient and researcher), are all validated and commonly used in experimental medicine studies.

The acceptability questionnaires relating to use of GP-ETB were created specifically for this study to obtain a data set for analysis of GP-ETB user satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and aged between 18 and 65 inclusive.
2. Diagnosed by GP with a depressive episode requiring treatment with citalopram (new or recurrent diagnosis).
3. Prescribed citalopram by GP for treatment of depression within past 3 days but has not yet started taking medication.
4. Is intending to start citalopram treatment within 2 days of Visit 1.
5. Fluent English speaker.
6. Has not consumed more than 4 units of alcohol in the 24 hours prior to Visit 1 and has not consumed any alcohol in the 8 hours prior to Visit 1.
7. Has not smoked tobacco in the 2 hours prior to completing the GP-ETB at Visit 1.
8. Has not consumed any beverages containing caffeine for 2 hours prior to completing the GPETB at Visit 1.
9. Has not consumed any psychoactive substances for 24 hours prior to Visit 1.
10. Willing and able to comply with study procedures, including treatment with citalopram and study prohibitions and restrictions.
11. Patient must have signed the informed consent form prior to the first study related procedure indicating they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Pregnant or breastfeeding, or planning to become pregnant during study, as determined through interview with patient.
2. Currently taking antidepressant medication.
3. Has taken antidepressant medication in the past 3 months.
4. Currently taking anti-psychotic or regular sedative medication, or is likely to require these during the study.
5. Regular (at least every week) use of recreational drugs including cannabis, as determined through interview with patient.
6. History of alcohol or substance dependence within the last 12 months from Visit 1, as assessed using standard screening questions.
7. Unlikely to be able to complete GP-ETB test.
8. Requires immediate referral to secondary care mental health services.
9. Is employed by the investigator or is related to the investigator
10. Currently taking part in a drug study or another device study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in Quick Inventory of Depressive Symptomology - Self Report (QIDS-SR) score from baseline (pre-dose of citalopram) to Day 28-42 post first dose of citalopram | Baseline (pre first dose of citalopram) to day 28-42 post first dose of citalopram)
  The QIDS-SR is a self report questionnaire and will be completed at baseline pre first dose of citalopram and at day 28-42 post first dose of citalopram. Scores will be compared.
Change in General Practitioner P1vital Oxford Emotional Test Battery (GP-ETB) scores from baseline (pre first dose of citalopram) to Visit 2 (7-9 days post first dose of citalopram) | Baseline (pre first dose of citalopram) to day 7-9 post first dose of citalopram)
  Patients will complete the GP-ETB tasks at baseline and 7-9 days post their first dose of citalopram and the scores compared.

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression rating Scale (MADRS) score from baseline (pre-dose of citalopram) to Day 28-42 post first dose of citalopram | Baseline (pre first dose of citalopram) to day 28-42 post first dose of citalopram)
  The MADRS interview will be conducted at baseline and again at the end of the study (day 28-42 post first dose of citalopram) and the scores compared.
Acceptability questionnaire results | The questionnaire will be completed at Day 28-42 post first dose of citalopram and will measure the participant's experience of the GP-ETB tests performed during the study
  All participants will complete an acceptability questionnaire about ease of use of the medical device.This visit occurs between Day 28 and day 42 after the first dose of citalopram taken by the patient. The data will be subjective text fields and Yes/No answers.
Adverse Events (AEs), Adverse Device Effects (ADEs) and device deficiencies will be recorded at each visit in the participant Case Report Form (CRF) | AEs will be collected per patient from the baseline visit (day 0), from the time the consent form is signed, until study end (28-42 days post first dose of citalopram) or patient withdrawal.
  Assessment of safety will be made through AE's, ADEs and device deficiencies recorded on the Case Report Form for the study first patient enrolled (June 2014) throughout the study until last patient last visit (January 2015). AEs or ADEs that have not resolved by the time a patient leaves the study will be followed up until resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Browning, MRCPsych, Principal Investigator — P1vital Limited
Locations (10):
- United Kingdom (10):
  - Cornerstone Practice, March, Cambridgeshire
  - Knowle House Surgery, Plymouth, Devon
  - Wareham Surgery, Wareham, Dorset
  - Oak Street Medical Centre, Norwich, Norfolk
  - The Surgery, Burnhope, Northumberland
  - Harbottle Surgery, Morpeth, Northumberland
  - Rosedale Surgery, Carlton Colville, Suffolk
  - Atherstone Surgery, Atherstone, Warwickshire
  - Sherbourne Medical Centre, Royal Leamington Spa, Warwickshire
  - Bradford Road Medical Centre, Trowbridge, Wiltshire

IPD SHARING:
Plan to Share IPD: No